CLINICAL TRIAL: NCT02552186
Title: Non-invasive Clinical Pectus Index as a Measurement of Severity in Pectus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00067521
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Pectus Excavatum
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pectus Excavatum Group (Active Comparator): The first group (PE Group) will consist of patients presenting to the All Children's Hospital Johns Hopkins Medicine (ACH JHM) Pediatric Surgery or Cardiac Surgery Clinics and the outpatient clinic system at Johns Hopkins Hospital for evaluation of pectus excavatum. Clinical measurements will be obtained using calipers.
  Interventions: Other: Caliper measurement
- Control Group (No Intervention): The second group (Control Group) will be age and gender matched patients presenting to the Radiology department of ACH JHM undergoing CT chest for indications other than chest wall deformity.

INTERVENTIONS:
Other: Caliper measurement — Clinical caliper measurements will be taken and used to calculate the Clinical PI
  Arms: Pectus Excavatum Group

SUMMARY:
Pectus excavatum (PE), the most common congenital chest wall deformity, requires surgical repair when the degree of deformity is severe. Currently, the Pectus Index (PI) is used to classify PE severity. Calculation of the PI requires cross-sectional imaging of the chest, usually with computed tomography (CT) or Magnetic Resonance Imaging (MRI), to obtain the necessary measurements. However, CT delivers a high dose of ionizing radiation, which carries cumulative long-term risks of malignancy and MRI can be costly. The purpose of this study is to develop a method whereby accurate chest wall measurements can be obtained to quantify PE severity without the need for cross-sectional imaging.

DETAILED DESCRIPTION:
This is a prospective study. The study population will consist of 2 groups. The first group (PE Group) will consist of patients presenting to the Johns Hopkins All Children's Hospital (JHACH) Pediatric Surgery or Cardiac Surgery Clinics and the outpatient clinic system at Johns Hopkins Hospital for evaluation of pectus excavatum. The second group (Control Group) will be age and gender matched patients presenting to the Radiology department of JHACH undergoing CT chest for indications other than chest wall deformity. Clinical caliper measurements will be taken and used to calculate the Clinical PI.

The steps to obtain the clinical caliper measurements are as follows: With the subject lying down, a ruler will be placed across the chest and a second ruler will be used to measure the depth at the deepest point of the sternum. The 2nd ruler will then be used to measure the height of the horizontal ruler to the bed on both sides. All measurements will be made on end expiration. With the subject standing, a measuring tape will be placed around the chest at the point of the deepest sternal depression. The sternum, spine and the bilateral lateral chest locations will be marked with temporary ink. The tape will be kept as level as possible. Chest calipers will be used to measure from deepest point of sternum to posterior midline, posterior midline to anterior chest and the transverse chest diameter. Each measurement will be taken at end expiration. The circumference of the chest will be recorded.

Each set of measurements will be taken by 2 independent members of the research team. Attempts will be made to record the amount of time it takes to obtain the measurements. Consent will be obtained to photograph the process for illustrative purposes. Every attempt will be made to conceal the patient's identity by excluding the face from the photograph. In instances where the face is not able to be excluded, the facial features will be blurred.

Clinical measurements may be recorded during routine medical care at the provider's discretion. However, these measurements will be considered research procedures for the purposes of this trial. A copy of the measurements will be placed in the medical chart of subjects evaluated for PE for the provider's future reference. Measurements obtained in the Control group will be strictly for the purposes of the research protocol. All subjects, regardless of group, will be provided standard of care for all other medical conditions.

All CT and MRI performed for both PE and Control groups will be reviewed and the PI will be determined by a single, blinded radiologist. The radiologist determining the PI may not be the interpreting radiologist and will have no responsibility to provide a comprehensive interpretation of the study. The PI as determined by the research radiologist will be recorded separately from the subject's EMR in a research file. Having a single, blinded radiologist determine the PI for the entire research cohort will allow for consistency in determining the PI, as this is the gold standard to which we are comparing our clinical measurements.

ELIGIBILITY:
Inclusion Criteria:

* Group A (PE Group): All patients evaluated in the ACH JHM Pediatric Surgery or Cardiac Surgery Clinics, as well as in the outpatient clinic system at Johns Hopkins Hospital, for surgical correction of Pectus Excavatum.
* Group B (Control Group): Age and gender matched patients who undergo chest CT at the ACH JHM Radiology Department for indications other than Pectus Excavatum.

Exclusion Criteria:

* None

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 199 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity of clinically-derived threshold versus CT/MRI-derived thresholds | 5 years
  Sensitivity refers to the ability of the test to correctly identify those patients with the disease.
Specificity of clinically-derived threshold versus CT/MRI-derived thresholds | 5 years
  Specificity refers to the ability of the test to correctly identify those patients without the disease.
Receiver operator characteristic curve of clinically-derived threshold versus CT/MRI-derived thresholds | 5 years
  plot of the true positive rate against the false positive rate for the different possible cutpoints of a diagnostic test.

SECONDARY OUTCOMES:
Correlation coefficient | 5 years
  statistical measure of the strength of the relationship between the relative movements of two variables.
Cohen's Kappa coefficient | 5 years
  a statistic which measures inter-rater agreement for qualitative (categorical) items. It
Agreement between Clinical Pectus Index (CPI) and Pectus Index (PI)-derived from CT or MRI | 5 years
  determine how well each measure identifies the outcome desired

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Chandler, MD, Principal Investigator — JHACH
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States